CLINICAL TRIAL: NCT04401956
Title: Comparison of the Tolerance of Spelt and Wheat Bread in Humans With Suspected NCWS Considering Different Manufacturing Processes of Bread
Brief Title: Bread Study: Comparison of the Tolerance of Spelt and Wheat Bread
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Principal Investigator, Stephan C. Bischoff, MD, Professor, Professor Dr. med., University of Hohenheim
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: ErnMed-Brot
Record Dates: First submitted 2020-05-14; First posted 2020-05-26 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Non-celiac Gluten Sensitivity; Wheat Intolerance
Keywords: Human Nutrition; NCWS; Spelt; Wheat Bread
MeSH Terms: interventions — Bread

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Gluten free bread with added gluten (Active Comparator): Bread will be eaten by the participants for 4 consecutive days.
  Interventions: Other: bread
- Gluten free bread with added FODMAPs (Active Comparator): Bread will be eaten by the participants for 4 consecutive days.
  Interventions: Other: bread
- Traditional manufactured wheat bread (Experimental): Bread will be eaten by the participants for 4 consecutive days.
  Interventions: Other: bread
- Traditional manufactured spelt bread (Experimental): Bread will be eaten by the participants for 4 consecutive days.
  Interventions: Other: bread
- Conventional manufactured wheat bread (Experimental): Bread will be eaten by the participants for 4 consecutive days.
  Interventions: Other: bread
- Conventional manufactured spelt bread (Experimental): Bread will be eaten by the participants for 4 consecutive days.
  Interventions: Other: bread

INTERVENTIONS:
Other: bread — Different types of bread

SUMMARY:
This project aims to verify the hypothesis that spelt products are more tolerable than bread wheat products in a target group of individuals with self-diagnosed wheat sensitivity. In addition, the influence of different manufacturing processes will be considered.

DETAILED DESCRIPTION:
Wheat cereals are known to be capable of triggering wheat allergy and celiac disease. The prevalence of both diseases is about 1%. Recently, another clinical entity was described, the non-celiac wheat sensitivity (NCWS). The origin and mechanisms of NCWS are unclear at present, but the existence of this new disease entity has been proven by double-blind placebo-controlled challenge tests. Three different grain components have been proposed as triggers of NCWS, gluten, α-amylase trypsin inhibitors or fermentable carbohydrates (FODMAPs).

It is reported that individuals with self-diagnosed NCWS quite often tolerate spelt products much better, even though spelt shows a higher gluten content than bread wheat products. Therefore, the question arises whether this putative spelt tolerance can be confirmed on an objective basis and whether the underlying molecular mechanisms can be elucidated. So far, human study addressing such questions are lacking.

This project aims to verify the hypothesis that spelt products are more tolerable than bread wheat products in a target group of individuals with self-diagnosed wheat sensitivity. In addition, the influence of different manufacturing processes on wheat sensitivity will be revealed.

For this purpose, the trial involves individuals with self-diagnosed wheat sensitivity and spelt tolerance. Six different kinds of bread will be tested, including 4 wheat and spelt breads, each of them produced following a traditional or a conventional way. Aim of this part is to objective bread wheat and spelt intolerance in a defined population. To find out whether FODMAPs or gluten affect the tolerance of bread, two additional breads will be tested, a gluten-free bread with added gluten and a gluten-free bread with added FODMAPs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 ≤70 years
* Signed declaration of consent
* Willingness to adhere to the prescribed diet for the duration of the study
* Subjective bread wheat intolerance
* No known spelled intolerance
* No acute or chronic gastrointestinal diseases (e.g. celiac disease / wheat allergy)
* No participation in another clinical trial (current or within the past 30 days)
* Gluten-containing diet at least 6 weeks before the start of the study

Exclusion Criteria:

* Taking intestinal therapeutics, antibiotics, immunosuppressants or similar
* Pregnancy / lactation
* Relevant violations of the nutritional protocol
* Occurrence of relevant diseases (possibly individual decision)
* Revocation of consent
* Accommodation in a clinic or similar facility based on an official or judicial order

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Change of IBS-SSS Total score | Study examinations are at baseline, after wash out phases (day 3, 10, 17, 24, 31, 38) and after bread intervention phases (day 7, 14, 21, 28, 35, 42).)
  IBS-SSS Total score will be collected with a questionnaire

SECONDARY OUTCOMES:
Extraintestinal Symptoms | Study examinations are at baseline, after wash out phases (day 3, 10, 17, 24, 31, 38) and after bread intervention phases (day 7, 14, 21, 28, 35, 42).)
  The study team will ask the participants for typical extraintestinal symptoms in NCWS like headache, foggy-mind, nausea, heartburn, exhaustion
Blood and fecal markers | Study examinations are at baseline and after bread intervention phases (day 7, 14, 21, 28, 35, 42).
  Change of blood- and fecal markers that will reveal inflammation or intestinal permeability (Anti-gliadin Immunglobulin G antibody, lipase, ferritin, zonulin, calprotectin and lactoferrin)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hohenheim, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: Undecided